CLINICAL TRIAL: NCT01883193
Title: Women First: Preconception Maternal Nutrition
Acronym: WF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Instituto de Nutricion de Centroamerica y Panama (INCAP) (Unknown); Kinshasa School of Public Health (Other); Jawaharlal Nehru Medical College (Other); Aga Khan University (Other); RTI International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-1672; OPP1055867 (Other Grant/Funding Number: Bill & Melinda Gates Foundation); U10HD076474-01 (NIH)
Record Dates: First submitted 2013-06-18; First posted 2013-06-21 (Estimated); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Maternal Malnutrition; Growth Failure; Mortality; Morbidity; Stunting
Keywords: preconception maternal nutrition; LBW; Length-for-age; maternal nutrition supplement; multi-micronutrient fortified lipid-based supplement; infant growth; low-resource settings
MeSH Terms: conditions — Failure to Thrive; Growth Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1: Preconception (Experimental): Arm 1 will commence the comprehensive maternal nutrition intervention at 3-7 months postpartum. Delivery of the intervention will be monitored biweekly by collection of empty and unused sachets of the lipid-based supplement (LNS), maternal report, and casual observation of household behavior. Arm 1 participants will be weighed monthly and Body Mass Index (BMI) calculated. If BMI <20 an additional energy supplement will be provided. Menstrual history will be obtained at each visit and a urine pregnancy test will be performed if menses is delayed.
  Interventions: Dietary Supplement: Comprehensive Maternal Nutrition Intervention
- Arm 2: Pregnancy (Experimental): Participants in Arm 2 will commence the same comprehensive maternal nutrition intervention at 12 weeks gestation.
  Interventions: Dietary Supplement: Comprehensive Maternal Nutrition Intervention
- Arm 3: Control (No Intervention): Participants in Arm 3 will receive biweekly visits to monitor pregnancy status. No health advice will be given other than information about prenatal care, location of delivery, and breastfeeding education in the third trimester.

INTERVENTIONS:
Dietary Supplement: Comprehensive Maternal Nutrition Intervention — The nutrition intervention will be delivered before conception or at 12 weeks gestation and continued through delivery and compared with a control group. The supplement to be used is a multi-micronutrient (MMN) fortified lipid-based supplement composed of dried skimmed milk, soybean and peanut extract, sugar, maltodextrin stabilizers, and emulsifiers.
  Other Names: multi micronutrient (MMN) fortified lipid-based supplement; lipid-based nutrient supplement; LNS
  Arms: Arm 1: Preconception; Arm 2: Pregnancy

SUMMARY:
Multi-country three-arm, individually randomized, non-masked, controlled trial to ascertain the benefits of ensuring optimal maternal nutrition before conception and providing an evidence base for programmatic priority directed to minimizing the risk of malnutrition in all females of reproductive age.

DETAILED DESCRIPTION:
The objective is to determine the benefits to the offspring of women in poor, food-insecure environments of commencing a daily comprehensive maternal nutrition supplement (with additional balanced calorie/protein supplement for underweight participants) ≥ 3 months prior to conception versus the benefits of commencing the same supplement at 12 weeks gestation and also to compare offspring outcomes with those of a control group which receives no supplement.

ELIGIBILITY:
Inclusion Criteria:

* 16-35 years of age;
* expectation to have first or further pregnancy without intent to utilize contraception
* Hb >8 g/dL

Exclusion Criteria:

* Nulliparous women who do not agree to hospital delivery (equipped for caesarian section) or/and do not have ready access to such a facility.

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7374 (Actual)
Dates: Start 2013-08; Primary Completion 2017-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Neonatal linear growth | <24 hours of age
  Research assistants will obtain neonatal length measurement at <24 hours of age.

SECONDARY OUTCOMES:
Length-for-age Z-scores | age 0.5, 1, 3, 6, 12, 18 and 24 months postnatal
  Research assistants will obtain infant anthropometry measurements, which include length, head circumference, triceps skin folds, Mid Upper Arm Circumference (MUAC), and weight, at age 0.5, 1, 3, 6, 12, 18 and 24 months of age. Length-for-age Z-scores will be compared for offspring of mothers randomized to the three intervention arms.
Estimate fetal growth | 12 weeks gestation
  Ultrasound measurements will be undertaken at 12 weeks gestation with the goals of confirming gestational age and estimating fetal growth.
Mean birth weight | at birth
  As a dichotomous variable, the cutoff of 2500 g does not have the power of the continuum of birth length, but is included because of the long history of use in determining which newborns are severely underweight and this association with impaired neonatal and long-term prognosis. The design of this study will allow distinction between pre-term birth (PTB) and growth retardation of the term infant (mature IUGR).
Incidence of low birth weight (LBW) infants | at birth
  As a dichotomous variable, the cutoff of 2500 g does not have the power of the continuum of birth length, but is included because of the long history of use in determining which newborns are severely underweight and this association with impaired neonatal and long-term prognosis. The design of this study will allow distinction between pre-term birth (PTB) and growth retardation of the term infant (mature IUGR).
Perinatal Mortality | From 20 weeks gestation through 1 month of age
  The outcome is to determine, in poor food insecure communities if a daily comprehensive maternal nutrition supplement starting ≥ 3 months preconception and continuing throughout pregnancy will reduce the incidence of offspring perinatal mortality (including still births), compared with that for offspring of mothers who commence the same supplement starting at 12-16 weeks gestation.
Incidence of severe neonatal and infant infectious disease | birth to 6 months of age
  Outcome measure is number of acute visits / admissions to health center/hospital for severe infectious disease. This secondary outcome will provide insight into the importance of maternal and fetal nutrition in the early prenatal development of host-defense mechanisms and, through comparison with the prenatal and control Arms, on the importance of maternal nutrition throughout pregnancy. It is further intended to collect minor morbidity data.
Epigenome (Maternal) | baseline, 12 and 34 weeks gestation, delivery, and 3 months postpartum (maternal); 2 weeks and 3 months of age (infant)
  To compare longitudinal changes between groups in the maternal epigenome (including blood, buccal swabs, and possibly other readily obtainable samples) at baseline, 12 weeks pregnancy (prior to initiation of LNS in Arm 2), 34 weeks pregnancy, and at 3 months postpartum. Also will collect placental, fetal and cord blood epigenome at delivery by group and infant epigenome at 3 months with fingerstick blood and buccal swabs.
Epigenome (Infant) | 2 weeks and 3 months of age
  To compare longitudinal changes between groups in the maternal epigenome (including blood, buccal swabs, and possibly other readily obtainable samples) at baseline, 12 weeks pregnancy (prior to initiation of LNS in Arm 2), 34 weeks pregnancy, and at 3 months postpartum. Also will collect placental, fetal and cord blood epigenome at delivery by group and infant epigenome at 3 months with fingerstick blood and buccal swabs.
Deep phenotyping of maternal metabolic and nutritional status | 12 and 34 weeks gestation, delivery, and 3 months postpartum
  The outcome represents deep phenotyping by measuring in maternal tissues: hormones, metabolites, measures of inflammation, oxidant stress and immune function/status, and nutrient biomarkers as possible indices of fundamental metabolic alterations resulting from improved long-term maternal nutrition in food insecure populations. Longitudinal blood samples will be collected from maternal participants in Arms 1 and 2 at baseline, 12 weeks gestation (prior to initiation of LNS in Arm 2), 34 weeks gestation, delivery and 3 months postpartum. Samples will also be collected from participants in Arm 3 at 34 weeks gestation and at 3 months postpartum.
Microbiome (maternal) | 12 & 34 weeks gestation and delivery (maternal)
  Based on potential long-term effects on maternal nutritional and metabolic state from preconception intervention, we hypothesize that the gut microbiota will differ between the two intervention arms at the three proposed time points.
Microbiome (infant) | 14 days and 3 months of age (infant)
  Based on potential long-term effects on maternal nutritional and metabolic state from preconception intervention, we hypothesize that the gut microbiota will differ between the two intervention arms at the three proposed time points.
Composition of breast milk | 14 days postpartum
  We hypothesize that improved maternal nutrition at the time of greatest plasticity in early pregnancy will favorably influence maternal metabolic and nutritional status throughout pregnancy and thus potentially the composition of breast milk in terms of hormonal content, immune factors, cytokines, and gut growth factors.
Neurodevelopment assessment | 24 mo age
  Offspring randomized to receive neurodevelopmental evaluation (BSID-III or InterNDA, 2:1 ratio) at 24 mo of age
Gestational weight gain (GWG) | Enrollment to delivery
  Describe GWG and its associations with fetal growth and birth outcomes within each country by baseline maternal nutritional status (BMI) and the receipt of nutrition interventions. Evaluate how GWG might mediate the effects of maternal nutrition interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Krebs, MD,MS, Principal Investigator — University of Colorado, Denver; Michael Hambidge, MD, SciD, Principal Investigator — University of Colorado, Denver
Locations (4):
- Kinshasa School of Public Health, Kinshasa, Democratic Republic of the Congo
- INCAP, Guatemala City, Guatemala
- Jawaharlal Nehru Medical College, Belagavi, India
- Aga Khan University, Karachi, Pakistan

REFERENCES:
- [Background] Hambidge KM, Krebs NF, Westcott JE, Garces A, Goudar SS, Kodkany BS, Pasha O, Tshefu A, Bose CL, Figueroa L, Goldenberg RL, Derman RJ, Friedman JE, Frank DN, McClure EM, Stolka K, Das A, Koso-Thomas M, Sundberg S; Preconception Trial Group. Preconception maternal nutrition: a multi-site randomized controlled trial. BMC Pregnancy Childbirth. 2014 Mar 20;14:111. doi: 10.1186/1471-2393-14-111. PMID 24650219
- [Background] Hambidge KM, Westcott JE, Garces A, Figueroa L, Goudar SS, Dhaded SM, Pasha O, Ali SA, Tshefu A, Lokangaka A, Derman RJ, Goldenberg RL, Bose CL, Bauserman M, Koso-Thomas M, Thorsten VR, Sridhar A, Stolka K, Das A, McClure EM, Krebs NF; Women First Preconception Trial Study Group. A multicountry randomized controlled trial of comprehensive maternal nutrition supplementation initiated before conception: the Women First trial. Am J Clin Nutr. 2019 Feb 1;109(2):457-469. doi: 10.1093/ajcn/nqy228. PMID 30721941
- [Background] Hambidge KM, Bann CM, McClure EM, Westcott JE, Garces A, Figueroa L, Goudar SS, Dhaded SM, Pasha O, Ali SA, Derman RJ, Goldenberg RL, Koso-Thomas M, Somannavar MS, Herekar V, Khan U, Krebs NF. Maternal Characteristics Affect Fetal Growth Response in the Women First Preconception Nutrition Trial. Nutrients. 2019 Oct 21;11(10):2534. doi: 10.3390/nu11102534. PMID 31640153
- [Background] Gilley SP, Weaver NE, Sticca EL, Jambal P, Palacios A, Kerns ME, Anand P, Kemp JF, Westcott JE, Figueroa L, Garces AL, Ali SA, Pasha O, Saleem S, Hambidge KM, Hendricks AE, Krebs NF, Borengasser SJ. Longitudinal Changes of One-Carbon Metabolites and Amino Acid Concentrations during Pregnancy in the Women First Maternal Nutrition Trial. Curr Dev Nutr. 2019 Nov 18;4(1):nzz132. doi: 10.1093/cdn/nzz132. eCollection 2020 Jan. PMID 32175519
- [Background] Lander RL, Hambidge KM, Westcott JE, Tejeda G, Diba TS, Mastiholi SC, Khan US, Garces A, Figueroa L, Tshefu A, Lokangaka A, Goudar SS, Somannavar MS, Ali SA, Saleem S, McClure EM, Krebs NF, Group OBOTWFPNT. Pregnant Women in Four Low-Middle Income Countries Have a High Prevalence of Inadequate Dietary Intakes That Are Improved by Dietary Diversity. Nutrients. 2019 Jul 10;11(7):1560. doi: 10.3390/nu11071560. PMID 31295916
- [Background] Krebs NF, Hambidge KM. Response to Editorial: Balancing the benefits of maternal nutritional interventions; time to put women first! Am J Clin Nutr. 2019 Aug 1;110(2):521-522. doi: 10.1093/ajcn/nqz077. No abstract available. PMID 31367762
- [Background] Borengasser SJ, Baker PR 2nd, Kerns ME, Miller LV, Palacios AP, Kemp JF, Westcott JE, Morrison SD, Hernandez TL, Garces A, Figueroa L, Friedman JE, Hambidge KM, Krebs NF. Preconception Micronutrient Supplementation Reduced Circulating Branched Chain Amino Acids at 12 Weeks Gestation in an Open Trial of Guatemalan Women Who Are Overweight or Obese. Nutrients. 2018 Sep 11;10(9):1282. doi: 10.3390/nu10091282. PMID 30208589
- [Background] Aziz Ali S, Abbasi Z, Feroz A, Hambidge KM, Krebs NF, Westcott JE, Saleem S. Factors associated with anemia among women of the reproductive age group in Thatta district: study protocol. Reprod Health. 2019 Mar 18;16(1):34. doi: 10.1186/s12978-019-0688-7. PMID 30885226
- [Background] Tang M, Frank DN, Tshefu A, Lokangaka A, Goudar SS, Dhaded SM, Somannavar MS, Hendricks AE, Ir D, Robertson CE, Kemp JF, Lander RL, Westcott JE, Hambidge KM, Krebs NF. Different Gut Microbial Profiles in Sub-Saharan African and South Asian Women of Childbearing Age Are Primarily Associated With Dietary Intakes. Front Microbiol. 2019 Aug 14;10:1848. doi: 10.3389/fmicb.2019.01848. eCollection 2019. PMID 31474951
- [Background] Ali SA, Khan U, Abrejo F, Saleem S, Hambidge MK, Krebs NF, Westcott JE, Goldenberg RL, McClure EM, Pasha O. Challenges of Implementing an Individual Randomized Controlled Trial (Women First: Preconception Maternal Nutrition Study) in a Rural Study Site: A Case Study From Pakistan. Nutr Metab Insights. 2019 Jul 4;21:1178638819852059. doi: 10.1177/1178638819852059. eCollection 2019. PMID 31320804
- [Background] Dhaded SM, Hambidge KM, Ali SA, Somannavar M, Saleem S, Pasha O, Khan U, Herekar V, Vernekar S, Kumar S Y, Westcott JE, Thorsten VR, Sridhar A, Das A, McClure E, Derman RJ, Goldenberg RL, Koso-Thomas M, Goudar SS, Krebs NF. Preconception nutrition intervention improved birth length and reduced stunting and wasting in newborns in South Asia: The Women First Randomized Controlled Trial. PLoS One. 2020 Jan 29;15(1):e0218960. doi: 10.1371/journal.pone.0218960. eCollection 2020. PMID 31995570
- [Background] Hambidge KM, Krebs NF, Garces A, Westcott JE, Figueroa L, Goudar SS, Dhaded S, Pasha O, Aziz Ali S, Tshefu A, Lokangaka A, Thorsten VR, Das A, Stolka K, McClure EM, Lander RL, Bose CL, Derman RJ, Goldenberg RL, Bauserman M. Anthropometric indices for non-pregnant women of childbearing age differ widely among four low-middle income populations. BMC Public Health. 2017 Jul 24;18(1):45. doi: 10.1186/s12889-017-4509-z. PMID 28738791
- [Background] Lander RL, Hambidge KM, Krebs NF, Westcott JE, Garces A, Figueroa L, Tejeda G, Lokangaka A, Diba TS, Somannavar MS, Honnayya R, Ali SA, Khan US, McClure EM, Thorsten VR, Stolka KB; Women First Preconception Nutrition Trial Group. Repeat 24-hour recalls and locally developed food composition databases: a feasible method to estimate dietary adequacy in a multi-site preconception maternal nutrition RCT. Food Nutr Res. 2017 Apr 11;61(1):1311185. doi: 10.1080/16546628.2017.1311185. eCollection 2017. PMID 28469549
- [Background] Krebs NF, Hambidge KM, Westcott JL, Garces AL, Figueroa L, Tsefu AK, Lokangaka AL, Goudar SS, Dhaded SM, Saleem S, Ali SA, Bose CL, Derman RJ, Goldenberg RL, Thorsten VR, Sridhar A, Chowdhury D, Das A; Women First Preconception Maternal Nutrition Study Group. Growth from Birth Through Six Months for Infants of Mothers in the "Women First" Preconception Maternal Nutrition Trial. J Pediatr. 2021 Feb;229:199-206.e4. doi: 10.1016/j.jpeds.2020.09.032. Epub 2020 Sep 18. PMID 32956698
- [Background] Ali SA, Abbasi Z, Shahid B, Moin G, Hambidge KM, Krebs NF, Westcott JE, McClure EM, Goldenberg RL, Saleem S. Prevalence and determinants of anemia among women of reproductive age in Thatta Pakistan: Findings from a cross-sectional study. PLoS One. 2020 Sep 24;15(9):e0239320. doi: 10.1371/journal.pone.0239320. eCollection 2020. PMID 32970719
- [Background] Aziz Ali S, Khan U, Abrejo F, Vollmer B, Saleem S, Hambidge KM, Krebs NF, Westcott JE, Goldenberg RL, McClure EM, Pasha O. Use of Smokeless Tobacco Before Conception and Its Relationship With Maternal and Fetal Outcomes of Pregnancy in Thatta, Pakistan: Findings From Women First Study. Nicotine Tob Res. 2021 Aug 4;23(8):1291-1299. doi: 10.1093/ntr/ntaa215. PMID 33084903
- [Derived] Gilley SP, Westcott JL, Kemp JF, Long JM, Hambidge KM, Shankar K, Krebs NF; Women First Trial Group. A Multicountry Analysis of Maternal Selenium Status in Pregnancy and Lactation and Infant Birth Outcomes: Findings from the Women First Maternal Preconception Study. J Nutr. 2025 Dec 27:101279. doi: 10.1016/j.tjnut.2025.101279. Online ahead of print. PMID 41461273
- [Derived] Ali SA, Valeri L, Kahe K, Genkinger JM, Saleem S, Jessani S, Goldenberg RL, Westcott JE, Kemp JF, Garces AL, Figueroa L, Goudar SS, Dhaded SM, Derman RJ, Tshefu A, Lokangaka AL, Bauserman MS, McClure EM, Koso Thomas M, Kuhn L, Krebs NF; Women First Preconception Nutrition Trial Group. Hemoglobin During Pregnancy Does Not Mediate the Relationship between Nutrition Supplements and Intrauterine Growth: A Secondary Data Analysis of Women First Preconception Nutrition Trial. J Nutr. 2025 Jul;155(7):2385-2397. doi: 10.1016/j.tjnut.2025.04.036. Epub 2025 May 19. PMID 40339908
- [Derived] Kemp JF, Hambidge KM, Westcott JL, Ali SA, Saleem S, Garces A, Figueroa L, Somannavar MS, Goudar SS, Long JM, Hendricks AE, Krebs NF; Women First Preconception Maternal Nutrition Trial Group. Zinc Supplementation Initiated Prior to or During Pregnancy Modestly Impacted Maternal Status and High Prevalence of Hypozincemia in Pregnancy and Lactation: The Women First Preconception Maternal Nutrition Trial. J Nutr. 2024 Jun;154(6):1917-1926. doi: 10.1016/j.tjnut.2024.04.018. Epub 2024 Apr 16. PMID 38621624
- [Derived] Fernandes M, Krebs NF, Westcott J, Tshefu A, Lokangaka A, Bauserman M, Garces AL, Figueroa L, Saleem S, Aziz SA, Goldenberg RL, Goudar SS, Dhaded SM, Derman RJ, Kemp JF, Koso-Thomas M, Sridhar A, M McClure E, Hambidge KM; Women First Preconception Nutrition Trial Study Group. Neurodevelopment, vision and auditory outcomes at age 2 years in offspring of participants in the 'Women First' maternal preconception nutrition randomised controlled trial. Arch Dis Child. 2023 Aug;108(8):622-631. doi: 10.1136/archdischild-2023-325352. Epub 2023 May 4. PMID 37142335
- [Derived] Krebs NF, Hambidge KM, Westcott JL, Garces AL, Figueroa L, Tshefu AK, Lokangaka AL, Goudar SS, Dhaded SM, Saleem S, Ali SA, Bauserman MS, Derman RJ, Goldenberg RL, Das A, Chowdhury D; Women First Preconception Maternal Nutrition Study Group. Birth length is the strongest predictor of linear growth status and stunting in the first 2 years of life after a preconception maternal nutrition intervention: the children of the Women First trial. Am J Clin Nutr. 2022 Jul 6;116(1):86-96. doi: 10.1093/ajcn/nqac051. PMID 35681255
- [Derived] Castillo-Castrejon M, Yang IV, Davidson EJ, Borengasser SJ, Jambal P, Westcott J, Kemp JF, Garces A, Ali SA, Saleem S, Goldenberg RL, Figueroa L, Hambidge KM, Krebs NF, Powell TL. Preconceptional Lipid-Based Nutrient Supplementation in 2 Low-Resource Countries Results in Distinctly Different IGF-1/mTOR Placental Responses. J Nutr. 2021 Mar 11;151(3):556-569. doi: 10.1093/jn/nxaa354. PMID 33382407